CLINICAL TRIAL: NCT04626583
Title: Safety of Locally Delivered Allogeneic Mesenchymal Stromal Cells for Promoting Corneal Repair
Brief Title: Safety of Locally Delivered Allogeneic Mesenchymal Stromal Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ali R Djalilian, Professor of Ophthalmology, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0334; W81XWH-18-1-0661 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-02

CONDITIONS: Mesenchymal Stromal Cells; Cornea; Safety; Corneal Defect
Keywords: Mesenchymal Stromal Cells; Corneal Defect
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Intervention Model Description: A longitudinal assessment using a classic dose-escalation study design to assess the safety of locally delivered allogenic mesenchymal stromal cells for promoting corneal repair.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose of allogeneic MSC (Active Comparator): Escalating doses of allogeneic MSC subconjunctival injection will be assigned 1,000,000 cells/50 µL at the low dose level.
  Interventions: Biological: Allogeneic MSC
- Medium dose of allogeneic MSC (Active Comparator): Escalating doses of allogeneic MSC subconjunctival injection will be assigned 3,000,000 cells/150 µL at the medium dose level.
  Interventions: Biological: Allogeneic MSC
- High dose of allogeneic MSC (Active Comparator): Escalating doses of allogeneic MSC subconjunctival injection will be assigned 6,000,000 cells total consisting of injection at 2 sites of 3,000,000 cells/150 µL each at the high dose level.
  Interventions: Biological: Allogeneic MSC

INTERVENTIONS:
Biological: Allogeneic MSC — Subconjunctival Injection of Allogeneic Mesenchymal Stromal Cells

SUMMARY:
This study is a longitudinal assessment using a classic dose-escalation study design to assess the safety and maximal tolerated dose (MTD) of locally delivered allogeneic mesenchymal stromal cells (MSC) for promoting corneal repair. The study will be conducted at Illinois Eye and Ear Infirmary located at University of Illinois at Chicago. The study will use digital conjunctival and corneal photography and corneal Scheimpflug Imaging, densitometry, and pachymetry for assessment of safety and corneal wound healing.

DETAILED DESCRIPTION:
The "Safety of Locally Delivered Allogeneic Mesenchymal Stem Cells for Promoting Corneal Repair Study" otherwise known as the "MSC Study," is designed to assess the safety of allogeneic bone marrow-derived MSC secreted factor on the ocular surface via subconjunctival injection of MSC, and also obtain a preliminary observation on the following:

1. Epithelial barrier integrity and/or wound closure.
2. Development of Scarring.
3. Final Visual Acuity.

The objective is to improve clinical outcomes in significant non-healing corneal wounds. To achieve these goals, the MSC Study will include a Phase I dose-escalation safety study.

ELIGIBILITY:
Inclusion Criteria:

Age:

• Patients 18 years of age or older

Visual Acuity:

• Best corrected distance visual acuity (BCDVA) score ≤ 75 ETDRS letters, (≥ 0.2 LogMAR, ≤ 20/32 Snellen or ≤ 0.625 decimal fraction) in the affected eye.

Ocular Health:

* Patients with moderate to severe chronic corneal epithelial disease in the setting of neurotrophic keratitis, limbal stem cell deficiency, or inflammatory dry eye disease.
* Epithelial disease refractory to all applicable standard / FDA approved non-surgical treatments (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops; anti-inflammatory therapy, and soft bandage contact lens).
* Evidence of impaired epithelial barrier manifested by fluorescein staining of the epithelium with a score 6 or higher by National Eye Institute grading.
* No objective clinical evidence of improvement since the last visit (≤50% reduction in fluorescein staining or ≤50% reduction in longest diameter of the epithelial defect).
* Patients with stage 1 (no epithelial defect) stage 2 (persistent epithelial defect, PED; without stromal loss) or stage 3 (corneal ulcer; with stromal loss) neurotrophic keratopathy 28-30 limited to ≤80% corneal diameter. Stromal loss in corneal ulcers cannot exceed 50%.
* Etiology of all persistent epithelial defects and corneal ulcers will be neurotrophic in nature. Neurotrophic keratopathy may be due to previous trauma such as chemical and thermal burns, systemic diseases like diabetes, post-infectious keratitis such as herpetic disease, or cranial nerve V palsies such as surgery for trigeminal neuralgia.
* PED or corneal ulceration refractory to one or more conventional non-surgical treatments (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops and medications that can decrease corneal sensitivity; therapeutic contact lenses).
* No objective clinical evidence of improvement in the PED or corneal ulceration within the week prior to study enrollment (e.g., ≤50% reduction in longest diameter in 1 week).
* Evidence of decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet aesthesiometer) within the area of the PED or corneal ulcer and outside of the area of the defect in at least one corneal quadrant.

Exclusion Criteria:

Visual Acuity:

• Patients with severe vision loss in the affected eye with no potential for visual improvement in the opinion of the investigator as a result of the study treatment.

Ocular Health:

* Any active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation not related to PED in the affected eye.
* History of any ocular surgery (including laser or refractive surgical procedures) in the affected eye within the three months before study enrollment. An exception to the preceding statement will be allowed if the ocular surgery is considered to be the cause of the PED. Ocular surgery in the affected eye will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period.
* Prior surgical procedure(s) for the treatment of a PED (e.g., complete tarsorrhaphy, conjunctival flap, etc.) in the affected eye with the exception of amniotic membrane transplantation. Patients previously treated with amniotic membrane transplantation may only be enrolled two weeks after the membrane has disappeared within the area of the PED or corneal ulcer or at least six weeks after the date of the amniotic membrane transplantation procedure. Patients previously treated with Botox (botulinum toxin) injections used to induce pharmacologic blepharoptosis are eligible for enrollment only if the last injection was given at least 90 days prior to enrollment in the study.
* Anticipated need for punctual occlusion during the study treatment period. Patients with punctual occlusion or punctual plugs inserted prior to the study are eligible for enrollment provided that the punctual occlusion is maintained during the study.
* Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting or perforation in the affected eye.
* Presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct (e.g., progressive or degenerative corneal or retinal conditions, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases).
* Any need for or anticipated change in the dose of systemic medications known to impair the function of the trigeminal nerve (e.g., neuroleptics, antipsychotic and antihistamine drugs). These treatments are allowed during the study if initiated prior to 30 days before study enrollment provided they remain stable throughout the course of the study treatment periods.

Study Procedures:

* Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein).
* History of drug, medication or alcohol abuse or addiction.
* Use of any investigational agent within 4 weeks of screening visit.
* Participation in another clinical study at the same time as the present study.
* Participants who are pregnant at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome: Incidence of treatment emergent adverse events (TEAE) assessed at 28 days. | Day #28
  Slit lamp exam will assess the safety of the treatment via TEAE at 28 days (participants will receive continued monitoring through 90 days). TEAE will be defined according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5) adverse event reference, and used to identify dose-limiting toxicity (DLT).
  The DLT will be defined as any non-corneal, ocular or systemic TEAE, with a Grade 2 toxicity without resolution after 14 days OR a Grade 3 toxicity, unless it can clearly be attributed to another cause. The DLT will be used to define the maximal tolerated dose (MTD).
  The MTD will be defined as the highest dose at which 0 to 1 of 6 patients experiences a dose-limiting toxicity (DLT). If a DLT occurs in 2 patients in a dosing cohort, then the MTD is considered exceeded and the dose will not be escalated.
Primary Efficacy Outcome: Proportion of participants with improvement in epithelial defect or barrier integrity relative to baseline (based on fluorescein staining) | Day #28
  Presence or absence of epithelial defect and epithelial staining grade following treatment, as determined by fluorescein staining observed via slit lamp examination, and photo-documented with digital corneal photography.

SECONDARY OUTCOMES:
Secondary Efficacy Outcomes: Visual Acuity | Enrollment, Treatment, and Days #1, #7, #14, #28, #90
  Best-corrected distance visual acuity will be measured using standard e-ETDRS protocols.
Secondary Efficacy Outcomes: Time to Completion of Corneal Epithelialization | Enrollment, Treatment, and Days #1, #7, #14, #28, #90
  Time to completion of corneal epithelialization will be assessed at each visit throughout the trial. Corneal epithelialization will be assessed as previously described.
Secondary Efficacy Outcomes: Durability of the Corneal Epithelialization and Healing | Enrollment, Treatment, and Days #1, #7, #14, #28, #90
  Durability of the corneal epithelization and healing will be assessed as an outcome measure at DAY #28 and DAY #90. Participants with corneal epithelialization prior to DAY #28 will be assessed at each subsequent follow-up visit (e.g., DAYS #7, #14, #28) to assess persistence of the healing response. Corneal epithelialization will be assessed as previously described.
Secondary Efficacy Outcomes: Corneal stromal haze | Enrollment and Days #7, #14, #28, #90
  Corneal stromal haze will be measured from Scheimpflug imaging and anterior segment OCT images (using Image J software). The treatment effect on corneal haze on DAY #28 will be compared relative to baseline.
Secondary Efficacy Outcomes: Corneal epithelial thickness | Enrollment and Days #7, #14, #28, #90
  Corneal epithelial thickness measured by anterior segment OCT imaging will assess the treatment effect on thickness on DAY #28 and compared relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Djalilian, MD, Principal Investigator — University of Illinois Chicago; Charlotte E Joslin, OD, PhD, Principal Investigator — University of Illinois Chicago
Locations (4):
- United States (4):
  - University of Illinois, Department of Ophthalmology and Visual Sciences, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Mass Eye and Ear Institute, Boston, Massachusetts
  - University of Pennsylvania Scheie Eye Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cockerham GC, Lemke S, Rice TA, Wang G, Glynn-Milley C, Zumhagen L, Cockerham KP. Closed-globe injuries of the ocular surface associated with combat blast exposure. Ophthalmology. 2014 Nov;121(11):2165-72. doi: 10.1016/j.ophtha.2014.06.009. Epub 2014 Aug 11. PMID 25124272
- [Background] Cockerham GC, Lemke S, Glynn-Milley C, Zumhagen L, Cockerham KP. Visual performance and the ocular surface in traumatic brain injury. Ocul Surf. 2013 Jan;11(1):25-34. doi: 10.1016/j.jtos.2012.09.004. Epub 2012 Oct 5. PMID 23321357
- [Background] Cockerham GC, Rice TA, Hewes EH, Cockerham KP, Lemke S, Wang G, Lin RC, Glynn-Milley C, Zumhagen L. Closed-eye ocular injuries in the Iraq and Afghanistan wars. N Engl J Med. 2011 Jun 2;364(22):2172-3. doi: 10.1056/NEJMc1010683. No abstract available. PMID 21631351
- [Background] Baradaran-Rafii A, Eslani M, Tseng SC. Sulfur mustard-induced ocular surface disorders. Ocul Surf. 2011 Jul;9(3):163-78. doi: 10.1016/s1542-0124(11)70026-x. PMID 21791191
- [Background] Baradaran-Rafii A, Eslani M, Haq Z, Shirzadeh E, Huvard MJ, Djalilian AR. Current and Upcoming Therapies for Ocular Surface Chemical Injuries. Ocul Surf. 2017 Jan;15(1):48-64. doi: 10.1016/j.jtos.2016.09.002. Epub 2016 Sep 17. PMID 27650263
- [Background] Eslani M, Baradaran-Rafii A, Movahedan A, Djalilian AR. The ocular surface chemical burns. J Ophthalmol. 2014;2014:196827. doi: 10.1155/2014/196827. Epub 2014 Jul 1. PMID 25105018
- [Background] Al-Moujahed A, Chodosh J. Outcomes of an algorithmic approach to treating mild ocular alkali burns. JAMA Ophthalmol. 2015 Oct;133(10):1214-6. doi: 10.1001/jamaophthalmol.2015.2302. No abstract available. PMID 26226389
- [Background] Prockop DJ, Oh JY. Mesenchymal stem/stromal cells (MSCs): role as guardians of inflammation. Mol Ther. 2012 Jan;20(1):14-20. doi: 10.1038/mt.2011.211. Epub 2011 Oct 18. PMID 22008910
- [Background] Mittal SK, Omoto M, Amouzegar A, Sahu A, Rezazadeh A, Katikireddy KR, Shah DI, Sahu SK, Chauhan SK. Restoration of Corneal Transparency by Mesenchymal Stem Cells. Stem Cell Reports. 2016 Oct 11;7(4):583-590. doi: 10.1016/j.stemcr.2016.09.001. Epub 2016 Sep 29. PMID 27693426
- [Background] Wang LT, Ting CH, Yen ML, Liu KJ, Sytwu HK, Wu KK, Yen BL. Human mesenchymal stem cells (MSCs) for treatment towards immune- and inflammation-mediated diseases: review of current clinical trials. J Biomed Sci. 2016 Nov 4;23(1):76. doi: 10.1186/s12929-016-0289-5. PMID 27809910
- [Background] Yun YI, Park SY, Lee HJ, Ko JH, Kim MK, Wee WR, Reger RL, Gregory CA, Choi H, Fulcher SF, Prockop DJ, Oh JY. Comparison of the anti-inflammatory effects of induced pluripotent stem cell-derived and bone marrow-derived mesenchymal stromal cells in a murine model of corneal injury. Cytotherapy. 2017 Jan;19(1):28-35. doi: 10.1016/j.jcyt.2016.10.007. Epub 2016 Nov 10. PMID 27840134
- [Background] Ye J, Yao K, Kim JC. Mesenchymal stem cell transplantation in a rabbit corneal alkali burn model: engraftment and involvement in wound healing. Eye (Lond). 2006 Apr;20(4):482-90. doi: 10.1038/sj.eye.6701913. PMID 15895027
- [Background] Yao L, Li ZR, Su WR, Li YP, Lin ML, Zhang WX, Liu Y, Wan Q, Liang D. Role of mesenchymal stem cells on cornea wound healing induced by acute alkali burn. PLoS One. 2012;7(2):e30842. doi: 10.1371/journal.pone.0030842. Epub 2012 Feb 17. PMID 22363499
- [Background] Roddy GW, Oh JY, Lee RH, Bartosh TJ, Ylostalo J, Coble K, Rosa RH Jr, Prockop DJ. Action at a distance: systemically administered adult stem/progenitor cells (MSCs) reduce inflammatory damage to the cornea without engraftment and primarily by secretion of TNF-alpha stimulated gene/protein 6. Stem Cells. 2011 Oct;29(10):1572-9. doi: 10.1002/stem.708. PMID 21837654
- [Background] Oh JY, Kim MK, Shin MS, Lee HJ, Ko JH, Wee WR, Lee JH. The anti-inflammatory and anti-angiogenic role of mesenchymal stem cells in corneal wound healing following chemical injury. Stem Cells. 2008 Apr;26(4):1047-55. doi: 10.1634/stemcells.2007-0737. Epub 2008 Jan 10. PMID 18192235
- [Background] Ma Y, Xu Y, Xiao Z, Yang W, Zhang C, Song E, Du Y, Li L. Reconstruction of chemically burned rat corneal surface by bone marrow-derived human mesenchymal stem cells. Stem Cells. 2006 Feb;24(2):315-21. doi: 10.1634/stemcells.2005-0046. Epub 2005 Aug 18. PMID 16109757
- [Background] Li F, Zhao SZ. Control of Cross Talk between Angiogenesis and Inflammation by Mesenchymal Stem Cells for the Treatment of Ocular Surface Diseases. Stem Cells Int. 2016;2016:7961816. doi: 10.1155/2016/7961816. Epub 2016 Mar 24. PMID 27110252
- [Background] Cejkova J, Trosan P, Cejka C, Lencova A, Zajicova A, Javorkova E, Kubinova S, Sykova E, Holan V. Suppression of alkali-induced oxidative injury in the cornea by mesenchymal stem cells growing on nanofiber scaffolds and transferred onto the damaged corneal surface. Exp Eye Res. 2013 Nov;116:312-23. doi: 10.1016/j.exer.2013.10.002. Epub 2013 Oct 18. PMID 24145108
- [Background] Bartlett RS, Guille JT, Chen X, Christensen MB, Wang SF, Thibeault SL. Mesenchymal stromal cell injection promotes vocal fold scar repair without long-term engraftment. Cytotherapy. 2016 Oct;18(10):1284-96. doi: 10.1016/j.jcyt.2016.07.005. PMID 27637759
- [Background] Bara JJ, Richards RG, Alini M, Stoddart MJ. Concise review: Bone marrow-derived mesenchymal stem cells change phenotype following in vitro culture: implications for basic research and the clinic. Stem Cells. 2014 Jul;32(7):1713-23. doi: 10.1002/stem.1649. PMID 24449458
- [Background] Ivy SP, Siu LL, Garrett-Mayer E, Rubinstein L. Approaches to phase 1 clinical trial design focused on safety, efficiency, and selected patient populations: a report from the clinical trial design task force of the national cancer institute investigational drug steering committee. Clin Cancer Res. 2010 Mar 15;16(6):1726-36. doi: 10.1158/1078-0432.CCR-09-1961. Epub 2010 Mar 9. PMID 20215542
- [Background] Ghazaryan E, Zhang Y, He Y, Liu X, Li Y, Xie J, Su G. Mesenchymal stem cells in corneal neovascularization: Comparison of different application routes. Mol Med Rep. 2016 Oct;14(4):3104-12. doi: 10.3892/mmr.2016.5621. Epub 2016 Aug 11. PMID 27514011
- [Background] Stevens S. Administering a subconjunctival injection. Community Eye Health. 2009 Mar;22(69):15. No abstract available. PMID 19506718
- [Background] Cook N, Hansen AR, Siu LL, Abdul Razak AR. Early phase clinical trials to identify optimal dosing and safety. Mol Oncol. 2015 May;9(5):997-1007. doi: 10.1016/j.molonc.2014.07.025. Epub 2014 Aug 14. PMID 25160636
- [Background] Sacchetti M, Lambiase A. Diagnosis and management of neurotrophic keratitis. Clin Ophthalmol. 2014 Mar 19;8:571-9. doi: 10.2147/OPTH.S45921. eCollection 2014. PMID 24672223
- [Background] Bonini S, Rama P, Olzi D, Lambiase A. Neurotrophic keratitis. Eye (Lond). 2003 Nov;17(8):989-95. doi: 10.1038/sj.eye.6700616. PMID 14631406
- [Background] Semeraro F, Forbice E, Romano V, Angi M, Romano MR, Filippelli ME, Di Iorio R, Costagliola C. Neurotrophic keratitis. Ophthalmologica. 2014;231(4):191-7. doi: 10.1159/000354380. Epub 2013 Oct 2. PMID 24107451
- [Background] Arnalich-Montiel F, Hernandez-Verdejo JL, Oblanca N, Munoz-Negrete FJ, De Miguel MP. Comparison of corneal haze and visual outcome in primary DSAEK versus DSAEK following failed DMEK. Graefes Arch Clin Exp Ophthalmol. 2013 Nov;251(11):2575-84. doi: 10.1007/s00417-013-2460-y. Epub 2013 Sep 6. PMID 24008847
- [Background] Elflein HM, Hofherr T, Berisha-Ramadani F, Weyer V, Lampe C, Beck M, Pitz S. Measuring corneal clouding in patients suffering from mucopolysaccharidosis with the Pentacam densitometry programme. Br J Ophthalmol. 2013 Jul;97(7):829-33. doi: 10.1136/bjophthalmol-2012-302913. Epub 2013 May 17. PMID 23685998
- [Background] Pahuja N, Shetty R, Subbiah P, Nagaraja H, Nuijts RM, Jayadev C. Corneal Densitometry: Repeatability in Eyes With Keratoconus and Postcollagen Cross-Linking. Cornea. 2016 Jun;35(6):833-7. doi: 10.1097/ICO.0000000000000800. PMID 27027920
- [Background] Akkaya Turhan S, Toker E. Changes in Corneal Density After Accelerated Corneal Collagen Cross-linking With Different Irradiation Intensities and Energy Exposures: 1-Year Follow-up. Cornea. 2017 Nov;36(11):1331-1335. doi: 10.1097/ICO.0000000000001362. PMID 28872519
- [Background] Enders P, Holtick U, Schaub F, Tuchscherer A, Hermann MM, Scheid C, Cursiefen C, Bachmann BO. Corneal Densitometry for Quantification of Corneal Deposits in Monoclonal Gammopathies. Cornea. 2017 Apr;36(4):470-475. doi: 10.1097/ICO.0000000000001078. PMID 27841786
- [Background] Gutierrez R, Lopez I, Villa-Collar C, Gonzalez-Meijome JM. Corneal transparency after cross-linking for keratoconus: 1-year follow-up. J Refract Surg. 2012 Nov;28(11):781-6. doi: 10.3928/1081597X-20121011-06. PMID 23347372
- [Background] Greenstein SA, Fry KL, Bhatt J, Hersh PS. Natural history of corneal haze after collagen crosslinking for keratoconus and corneal ectasia: Scheimpflug and biomicroscopic analysis. J Cataract Refract Surg. 2010 Dec;36(12):2105-14. doi: 10.1016/j.jcrs.2010.06.067. PMID 21111314
- [Background] Weiner X, Baumeister M, Kohnen T, Buhren J. Repeatability of lens densitometry using Scheimpflug imaging. J Cataract Refract Surg. 2014 May;40(5):756-63. doi: 10.1016/j.jcrs.2013.10.039. PMID 24767909
- [Background] Kim BZ, Jordan CA, McGhee CN, Patel DV. Natural history of corneal haze after corneal collagen crosslinking in keratoconus using Scheimpflug analysis. J Cataract Refract Surg. 2016 Jul;42(7):1053-9. doi: 10.1016/j.jcrs.2016.04.019. PMID 27492105
- [Background] Boulze-Pankert M, Dariel R, Hoffart L. Corneal Scheimpflug Densitometry Following Photorefractive Keratectomy in Myopic Eyes. J Refract Surg. 2016 Nov 1;32(11):788-791. doi: 10.3928/1081597X-20160720-02. PMID 27824385
- [Background] McLaren JW, Wacker K, Kane KM, Patel SV. Measuring Corneal Haze by Using Scheimpflug Photography and Confocal Microscopy. Invest Ophthalmol Vis Sci. 2016 Jan 1;57(1):227-35. doi: 10.1167/iovs.15-17657. PMID 26803798
- See also: Considerations for the Design of Early-Phase Clinical Trials of Cellular and Gene Therapy Products — https://www.fda.gov/media/106369/download